CLINICAL TRIAL: NCT01095731
Title: Phase II Study of the Effects of Tiopronin on 3-Aminopropanal Level & Neurologic Outcome After Aneurysmal Subarachnoid Hemorrhage
Brief Title: The Effects of Tiopronin on 3-Aminopropanal Level & Neurologic Outcome After Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: E. Sander Connolly (Other)
Collaborators: University of Florida (Other); University of Washington (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, E. Sander Connolly, Professor of Neurological Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAA8597; 1R01FD003728-01 (FDA)
Record Dates: First submitted 2010-03-25; First posted 2010-03-30 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aneurysm; aneurysmal; subarachnoid; hemorrhage; haemorrhage; neuroprotection; 3-aminopropanal; 3AP; polyamine oxidase; spermine; spermidine; vasospasm; cerebral ischemia; neurosurgery; neurological intensive care unit; NICU; Tiopronin; Thiola; FDA; Thiopronin; Thiosol; Tioglis; Acadione; Capen; Captimer; Epatiol; Vincol; Mucolysin; Sutilan; Meprin; Thiolpropionamidoacetic acid; Mercaptopropionyl glycine; 2 MPG
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Hemorrhage; Brain Ischemia | interventions — Tiopronin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill, Hunt Hess Grade I-V (Placebo Comparator): Good Grade (Hunt Hess I-III) and Poor Grade (Hunt Hess IV-V)
  Interventions: Drug: Placebo
- Tiopronin, Hunt Hess Grade I-V (Experimental): Good Grade (Hunt Hess I-III) and Poor Grade (Hunt Hess IV-V)
  Interventions: Drug: Tiopronin

INTERVENTIONS:
Drug: Tiopronin — Dosage will be 1 gram, 3 times daily. Drug dosing will be initiated at time of aSAH confirmation, for a length of 14 days or at hospital discharge.
  Other Names: IUPAC Name:2-(2-sulfanylpropanoylamino)acetic acid; CAS Number: 1953-02-2; Thiola; Thiopronin; Thiosol; Tioglis; Acadione; Capen; Captimer; Epatiol; Vincol; Mucolysin; Sutilan; Meprin (detoxicant); Thiolpropionamidoacetic acid; N-2-Mercaptopropionyl glycine; 2-(2-sulfanylpropanoylamino)ethanoic acid; 2-(2-sulfanylpropanoylamino)acetic acid
  Arms: Tiopronin, Hunt Hess Grade I-V
Drug: Placebo — Dosage will be 1 gram, 3 times daily. Drug dosing will be initiated at time of aSAH confirmation, for a length of 14 days or at hospital discharge.
  Other Names: placebo, sugar pill
  Arms: Sugar Pill, Hunt Hess Grade I-V

SUMMARY:
The purpose of this phase II study is to further assess the safety of tiopronin in aneurysmal subarachnoid hemorrhage(aSAH) patients in order to obtain preliminary data on the efficacy of tiopronin versus placebo in reducing serum and cerebrospinal fluid (CSF) 3AP levels in this patient population.

Funding Source - FDA Office of Orphan Products Development

DETAILED DESCRIPTION:
The annual rate of aSAH in United States is approximately 18 to 24 thousand cases each year. Mortality rates following aSAH range from 30-70% with 10-20% of survivors experiencing severe neurological disability. Following aSAH, a major cause of morbidity and mortality is vasospasm, which causes delayed ischemic neurologic deterioration. There is currently no effective treatment for preventing or ameliorating the damage that occurs following cerebral ischemia. A myriad of neuro-toxins are produced in the ischemic brain resulting in a vicious cycle of cellular death and destruction. The polyamines spermine and spermidine are metabolized by polyamine oxidase (PAO) into putrescine and 3-aminopropanal (3AP).

Tiopronin (Thiola) is an FDA approved drug used for the treatment of cystine stones in patients with cystinuria in the U.S. In Europe, it is also used for the treatment of rheumatoid arthritis and bronchial hypersecretion. In previous animal studies, we demonstrated that tiopronin is able to bind and neutralize the toxic effects of 3AP. We have shown in previous studies that aSAH patients have elevated 3AP levels, and higher levels correlate to a poor neurologic outcome.

The goals of this phase II multicenter, randomized, double-blinded safety and efficacy trial are to (1) further evaluate the safety of the drug in our patient population at the dose established in phase I; (2) demonstrate that tiopronin crosses the blood-brain barrier; (3) show that both serum and CSF 3AP levels are reduced by administration of tiopronin; and (4) demonstrate that a reduction in 3AP levels is associated with improved neurologic outcome in aSAH patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a recruiting center with aneurysmal subarachnoid hemorrhage
* Ability to initiate study drug treatment within 96 hours of aSAH onset.
* Ability to provide either informed or surrogate consent

Exclusion Criteria:

* Hypersensitivity to penicillamine
* Creatinine level greater than 1.5/mm^3 on admission
* Platelet count of less than 100,000/mm^3 on admission
* White blood cell count of less than 3.5/mm^3 on admission
* AST or ALT of greater than 60/L on admission or history of liver failure
* Pregnancy
* History of lupus, Goodpasture's syndrome, myasthenia gravis, pemphigus, nephrotic syndrome, glomerulonephritis, or renal failure
* Patients considered unable to comply with the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E Sander Connolly, M.D., Principal Investigator — Columbia University; Brian Hoh, M.D., Principal Investigator — University of Florida; Louis Kim, M.D., Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Columbia University Medical Center, New York, New York
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Linn FH, Rinkel GJ, Algra A, van Gijn J. Incidence of subarachnoid hemorrhage: role of region, year, and rate of computed tomography: a meta-analysis. Stroke. 1996 Apr;27(4):625-9. doi: 10.1161/01.str.27.4.625. PMID 8614919
- [Background] Hop JW, Rinkel GJ, Algra A, van Gijn J. Case-fatality rates and functional outcome after subarachnoid hemorrhage: a systematic review. Stroke. 1997 Mar;28(3):660-4. doi: 10.1161/01.str.28.3.660. PMID 9056628
- [Background] Mayer S, Kreiter K. Quality of life after subarachnoid hemorrhage. J Neurosurg. 2002 Sep;97(3):741-2; author reply 742. doi: 10.3171/jns.2002.97.3.0741. No abstract available. PMID 12296671
- [Background] Kassell NF, Sasaki T, Colohan AR, Nazar G. Cerebral vasospasm following aneurysmal subarachnoid hemorrhage. Stroke. 1985 Jul-Aug;16(4):562-72. doi: 10.1161/01.str.16.4.562. PMID 3895589
- [Background] Solenski NJ, Haley EC Jr, Kassell NF, Kongable G, Germanson T, Truskowski L, Torner JC. Medical complications of aneurysmal subarachnoid hemorrhage: a report of the multicenter, cooperative aneurysm study. Participants of the Multicenter Cooperative Aneurysm Study. Crit Care Med. 1995 Jun;23(6):1007-17. doi: 10.1097/00003246-199506000-00004. PMID 7774210
- [Background] Shohami E, Nates JL, Glantz L, Trembovler V, Shapira Y, Bachrach U. Changes in brain polyamine levels following head injury. Exp Neurol. 1992 Aug;117(2):189-95. doi: 10.1016/0014-4886(92)90126-b. PMID 1499692
- [Background] Ivanova S, Botchkina GI, Al-Abed Y, Meistrell M 3rd, Batliwalla F, Dubinsky JM, Iadecola C, Wang H, Gregersen PK, Eaton JW, Tracey KJ. Cerebral ischemia enhances polyamine oxidation: identification of enzymatically formed 3-aminopropanal as an endogenous mediator of neuronal and glial cell death. J Exp Med. 1998 Jul 20;188(2):327-40. doi: 10.1084/jem.188.2.327. PMID 9670045
- [Background] Dogan A, Rao AM, Hatcher J, Rao VL, Baskaya MK, Dempsey RJ. Effects of MDL 72527, a specific inhibitor of polyamine oxidase, on brain edema, ischemic injury volume, and tissue polyamine levels in rats after temporary middle cerebral artery occlusion. J Neurochem. 1999 Feb;72(2):765-70. doi: 10.1046/j.1471-4159.1999.0720765.x. PMID 9930751
- [Background] Seiler N. Polyamine oxidase, properties and functions. Prog Brain Res. 1995;106:333-44. doi: 10.1016/s0079-6123(08)61229-7. PMID 8584670
- [Background] Ivanova S, Batliwalla F, Mocco J, Kiss S, Huang J, Mack W, Coon A, Eaton JW, Al-Abed Y, Gregersen PK, Shohami E, Connolly ES Jr, Tracey KJ. Neuroprotection in cerebral ischemia by neutralization of 3-aminopropanal. Proc Natl Acad Sci U S A. 2002 Apr 16;99(8):5579-84. doi: 10.1073/pnas.082609299. Epub 2002 Apr 9. PMID 11943872
- [Background] Cockroft KM, Meistrell M 3rd, Zimmerman GA, Risucci D, Bloom O, Cerami A, Tracey KJ. Cerebroprotective effects of aminoguanidine in a rodent model of stroke. Stroke. 1996 Aug;27(8):1393-8. doi: 10.1161/01.str.27.8.1393. PMID 8711808
- [Background] Wood PL, Khan MA, Moskal JR. Neurochemical analysis of amino acids, polyamines and carboxylic acids: GC-MS quantitation of tBDMS derivatives using ammonia positive chemical ionization. J Chromatogr B Analyt Technol Biomed Life Sci. 2006 Feb 2;831(1-2):313-9. doi: 10.1016/j.jchromb.2005.12.031. Epub 2006 Jan 10. PMID 16406747
- [Background] Wood PL, Khan MA, Moskal JR, Todd KG, Tanay VA, Baker G. Aldehyde load in ischemia-reperfusion brain injury: neuroprotection by neutralization of reactive aldehydes with phenelzine. Brain Res. 2006 Nov 29;1122(1):184-90. doi: 10.1016/j.brainres.2006.09.003. Epub 2006 Oct 5. PMID 17026969
- [Background] Fisher CM, Kistler JP, Davis JM. Relation of cerebral vasospasm to subarachnoid hemorrhage visualized by computerized tomographic scanning. Neurosurgery. 1980 Jan;6(1):1-9. doi: 10.1227/00006123-198001000-00001. PMID 7354892
- [Background] Lindell A, Denneberg T, Hellgren E, Jeppsson JO, Tiselius HG. Clinical course and cystine stone formation during tiopronin treatment. Urol Res. 1995;23(2):111-7. doi: 10.1007/BF00307941. PMID 7676533
- [Derived] Ironside N, Christophe B, Bruce S, Carpenter AM, Robison T, Yoh N, Cremers S, Landry D, Frey HP, Chen CJ, Hoh BL, Kim LJ, Claassen J, Connolly ES. A phase II randomized controlled trial of tiopronin for aneurysmal subarachnoid hemorrhage. J Neurosurg. 2019 Jul 12;133(2):351-359. doi: 10.3171/2019.4.JNS19478. Print 2020 Aug 1. PMID 31299655
- See also: The Columbia University Medical Center Department of Neurosurgery Website — http://www.columbianeurosurgery.org/
- See also: The University of Florida Department of Neurosurgery Website — http://www.neurosurgery.ufl.edu/
- See also: The University of Washington Department of Neurosurgery Website — http://depts.washington.edu/neurosur/
- See also: Principle Investigator: E. Sander Connolly Jr. — http://www.columbianeurosurgery.org/doctors/e-sander-connolly-jr/
- See also: Connolly Cerebrovascular Research Laboratory — http://www.columbianeurosurgery.org/research/research-laboratories/cerebrovascular-research-laboratory/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants enrolled and one withdrew consent prior to randomization, resulting in allocation of 59 participants.
Period: Overall Study
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Started | 30 | 29
Completed | 29 | 27
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Customized [Count of Participants; unit: Participants]
  40 - 80 years | 30 | 29 | 59
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 12 | 5 | 17
  Unknown/Not reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 19 | 32
  Black | 5 | 3 | 8
  Asian | 1 | 0 | 1
  Hispanic | 8 | 4 | 12
  Other | 2 | 1 | 3
  Unknown/Not reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59
Diabetes Mellitus [Count of Participants; unit: Participants] | 3 | 3 | 6
Smoker [Count of Participants; unit: Participants] | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Cerebrospinal Fluid 3-aminopropanal (CSF-3AP) Levels
Description: The level of 3-aminopropanal (3-AP) in cerebrospinal fluid (CSF) measured in nmol/mL. CSF samples taken as a standard of care.
Time Frame: Day 7
Population: CSF samples were successfully collected on day 7 in 12 and 13 participants in the tiopronin and sugar pill arms, respectively.
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 12 | 13
nmol/mL | 11.1 (11.8) | 12.9 (17.6)

2. Secondary Outcome: Cerebrospinal Fluid 3-aminopropanal (CSF-3AP) Levels
Description: as for outcome 1
Time Frame: Day 14
Population: CSF samples were successfully collected on day 14 in 13 and 9 participants in the tiopronin and sugar pill arms respectively.
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 13 | 9
nmol/mL | 14.7 (18.8) | 9.9 (10.3)

3. Secondary Outcome: Modified Rankin Score (mRS) at Discharge
Description: The Modified Rankin Score (mRS) is a disability scale with possible scores ranging from 0 (no symptoms) to 5 (severe disability).
Time Frame: At time of discharge, approximately Day 14
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 29 | 27
score on a scale | 4 [2 to 5] | 4 [3 to 5]

4. Secondary Outcome: Modified Rankin Score (mRS) at 3 Months
Description: as for outcome 3
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 29 | 27
score on a scale | 3 [2 to 4] | 2 [1 to 4]

5. Secondary Outcome: Modified Rankin Score (mRS) at 12 Months
Description: as for outcome 3
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 29 | 27
score on a scale | 2 [1 to 2] | 2 [1 to 3]

6. Secondary Outcome: Barthel Index at Discharge
Description: Barthel index is a scale used to measure dependency in performing daily activities. Scores range from 0 (total dependency) to 100 (no dependency). A higher score indicates a better outcome.
Time Frame: At time of discharge, approximately Day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 29 | 27
score on a scale | 37 (53) | 30 (38)

7. Secondary Outcome: Barthel Index at 3 Months
Description: as for outcome 6
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 29 | 27
score on a scale | 83 (33) | 85 (28)

8. Secondary Outcome: Barthel Index at 12 Months
Description: as for outcome 6
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
Number analyzed (Participants) | 29 | 27
score on a scale | 94 (24) | 98 (5)

ADVERSE EVENTS:
Arm/Group | Tiopronin, Hunt Hess Grade I-V | Sugar Pill, Hunt Hess Grade I-V
All-Cause Mortality (participants affected / at risk) | 4/29 | 3/27
Serious Adverse Events (participants affected / at risk) | 6/29 | 9/27
Other Adverse Events (participants affected / at risk) | 13/29 | 16/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiopronin, Hunt Hess Grade I-V (N=29) | Sugar Pill, Hunt Hess Grade I-V (N=27)
Terminal Extubation (withdrawal of care) (General disorders) | 2 | 1
Ventriculitis (Nervous system disorders) | 1 | 0
Hypoxia (General disorders) | 1 | 0
Cardiopulmonary Arrest (General disorders) | 0 | 2
Neurological Deterioration (Nervous system disorders) | 1 | 1
Acidosis (General disorders) | 0 | 1
Staphylococcus aureus Infection (Infections and infestations) | 0 | 1
Fever (General disorders) | 1 | 0
Prolonged Intubation (General disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Fever of unknown origin (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiopronin, Hunt Hess Grade I-V (N=29) | Sugar Pill, Hunt Hess Grade I-V (N=27)
Fever (General disorders) | 5 | 5
Thrombosis (Vascular disorders) | 1 | 1
Seizure (Nervous system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Hypernatremia (General disorders) | 2 | 1
Hyponatremia (General disorders) | 3 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Leukopenia (Immune system disorders) | 1 | 0
Laryngeal edema (General disorders) | 1 | 0
Rash (General disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Arrhythmia (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No